CLINICAL TRIAL: NCT03528083
Title: Pediatric Bronchiolitis Quality Improvement to Reduce Unnecessary Use of Diagnostic Testing and Treatment
Brief Title: Pediatric Bronchiolitis Quality Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1219188
Record Dates: First submitted 2018-04-09; First posted 2018-05-17 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Children; Hospital
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a quality improvement process for all children diagnosed with bronchiolitis at our hospital who meet inclusion criteria. Outcomes for these patients will be compared with retrospective controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrospective Controls (No Intervention): A retrospective control group of patients with a diagnosis of bronchiolitis and meeting inclusion criteria will be used as a comparison group. These patients received usual care for bronchiolitis at our institution.
- Quality Improvement (Experimental): All patients diagnosed with bronchiolitis and meeting inclusion criteria will undergo the intervention of a bronchiolitis quality improvement process to improve bronchiolitis care quality at our institution.
  Interventions: Other: Bronchiolitis quality improvement

INTERVENTIONS:
Other: Bronchiolitis quality improvement — Patients in the intervention group will undergo a quality improvement process to improve care quality for bronchiolitis at our hospital.
  Arms: Quality Improvement

SUMMARY:
Bronchiolitis is a respiratory illness characterized by acute inflammation of the airways, typically caused by a virus. By definition, it impacts children between 2 months and 2 years of age and is the most common cause of hospitalization among infants in the first year of life (American Academy of Pediatrics). Children with this illness may exhibit respiratory distress, as well as symptoms of viral respiratory illness, such as sneezing, nasal congestion, and cough. Often, hospitalization is required for respiratory distress and to support hydration needs.

Evidence based guidelines for the treatment of acute viral bronchiolitis primarily involve supportive care, which most often includes supplemental oxygen, hydration, and suctioning of secretions. However, in practice, bronchiolitis care is highly variable, often involving therapies such as inhaled bronchodilators, systemic corticosteroids, inhaled hypertonic saline, continuous pulse oximetry, chest physiotherapy, antibacterial medications, and use of intravenous fluids, all of which have been shown to be unnecessary and costly. Unnecessary care remains although multiple published quality improvement studies centered on acute bronchiolitis have proven successful. Quality improvement interventions have shown reduced use of unnecessary treatments and reduced resource allocation. Therefore, the investigators will conduct a quality improvement process to improve adherence to bronchiolitis treatment guidelines for children with bronchiolitis treated at University of California Davis Children's Hospital.

DETAILED DESCRIPTION:
A multidisciplinary team, involving pediatric hospitalists, pediatric emergency physicians, residents, medical students, nurses and nurse managers, and respiratory therapists will be assembled. The investigators will participate in a value stream mapping process, to map out the current pediatric bronchiolitis care process and identify areas for improvement in efficiency and effectiveness. The investigators will then begin the iterative process of implementing improvements to the bronchiolitis care process. Interventions will be evidence-based and designed to improve compliance with bronchiolitis care guidelines, as set forth by the American Academy of Pediatrics. Examples of possible interventions may include creation of a bronchiolitis admission order set, implementation of an evidence-based bronchiolitis clinical pathway, and/or institution of standardized bronchiolitis discharge criteria. Interventions will be implemented in a stepwise fashion, utilizing successive plan-do-study-act cycles, with a minimum 2 month period between interventions to monitor outcomes. The investigators will track utilization of diagnostic testing and treatments within our intervention group, as compared to historical controls who also meet inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 2 years of age admitted to UC Davis Children's Hospital with any diagnosis of bronchiolitis

Exclusion Criteria:

* Children or adults greater than 2 years of age
* Children born at less than 35 weeks gestational age
* Children with underlying illnesses, such as chronic lung disease, congenital heart disease, other congenital anomalies including airway anomalies, or immunodeficiencies

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1321 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Chest x-ray utilization | Through study completion, an average of 19 months
  Percentage of patients meeting inclusion criteria who received a chest x-ray
Antibiotic utilization | Through study completion, an average of 19 months
  Percentage of patients meeting inclusion criteria who received antibiotics
Bronchodilator utilization | Through study completion, an average of 19 months
  Percentage of patients meeting inclusion criteria who received bronchodilators
Steroid utilization | Through study completion, an average of 19 months
  Percentage of patients meeting inclusion criteria who received steroids
Hypertonic saline utilization | Through study completion, an average of 19 months
  Percentage of patients meeting inclusion criteria who received nebulized hypertonic saline.
Chest physiotherapy utilization | Through study completion, an average of 19 months
  Percentage of patients meeting inclusion criteria who received chest physiotherapy
Intravenous fluid utilization | Through study completion, an average of 19 months
  Percentage of patients meeting inclusion criteria who received intravenous fluid
Continuous pulse oximetry utilization | Through study completion, an average of 19 months
  Percentage of patients meeting inclusion criteria who received continuous pulse oximetry
Supplemental oxygen utilization | Through study completion, an average of 19 months
  Percentage of patients meeting inclusion criteria who received supplemental oxygen

SECONDARY OUTCOMES:
Length of stay index | Through study completion, an average of 19 months
  A ratio of observed to expected length of stay for patients admitted with bronchiolitis, as compared to national standards
Readmission rate | Within 30 days following the index hospitalization discharge date
  Same hospital readmission rate for patients with a diagnosis of bronchiolitis
Emergency room revisit rate | Within 30 days following the index hospitalization discharge date
  Same hospital emergency room revisit rate for patients with a diagnosis of bronchiolitis
Bronchiolitis specific discharge instructions | Through study completion, an average of 19 months
  Percentage of patients meeting inclusion criteria who received bronchiolitis specific handout containing care instructions on discharge
Timely completion of discharge summary | Within 48 hours of discharge from the index hospitalization
  Percentage of patients meeting inclusion criteria who had a discharge summary completed
Timely routing of discharge summary | Within 48 hours of discharge from the index hospitalization
  Percentage of patients meeting inclusion criteria who had a discharge summary routed to their primary care provider
CC capture rate | Through study completion, an average of 19 months
  The capture rate for comorbid conditions within our charting for patients diagnosed with bronchiolitis
MCC capture rate | Through study completion, an average of 19 months
  The capture rate for major comorbid conditions within our charting for patients diagnosed with bronchiolitis

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hamline, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC David Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as data will be collected and reported in aggregate.